CLINICAL TRIAL: NCT07371819
Title: Effect of Saccharomyces Boulardii CNCM I-745 (Sb) on Bloody Diarrhea in Children. A Double Blind, Randomized, Controlled Study
Brief Title: Effect of Saccharomyces Boulardii CNCM I-745 (Sb) on Bloody Diarrhea in Children. A Double Blind, Randomized, Controlled Study ( Sb192-SUH )
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Hospital de Pediatría Prof. Dr. Juan P. Garrahan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Sb192-SUH
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Acute Bloody Diarrhea of 7 Days or Less Duration
Keywords: ACUTE BLOODY DIARRHEA. SACCHAROMYCES BOULARDII

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental)
  Interventions: Drug: Saccharomyces boulardi (Sb)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saccharomyces boulardi (Sb) — Drug: Saccharomyces Boulardii 250 MG Saccharomyces boulardi (Sb) 250 mg dose to be administered to the patient : - twice a day, to children from older than 1.0 year, up to 5.99 years, - or once a day to children 1year old or younger
  Arms: Treatment Arm
Drug: Placebo — Drug: Placebo Placebo to be administered to the patient : -twice a day, to children from older than 1.0 year, up to 5.99 years, - or once a day to children 1year old or younger
  Arms: Placebo

SUMMARY:
Acute diarrhea (AD) is one of the commonest illnesses in children. A particularly severe form of diarrhea is bloody diarrhea (BD).

Saccharomyces boulardii CNCM I-745 is a probiotic with demonstrated efficacy in children with acute diarrhea; however, evidence regarding its use in bloody diarrhea (BD) is lacking. This project aims to assess the efficacy and safety of Saccharomyces boulardii CNCM I-745 on bloody diarrhea in children.

The study objective are :

• To assess the efficacy of Sacharomyces Boulardi (SB) on acute bloody diarrhea in children aged 0 - 5 years. Indicators: duration of bloody diarrhea, daily frequency of stools with blood, daily frequency of total stools with or without blood during follow up.

• To assess the most frequent bacterial agents

• To assess the safety of the product. The study is a double blind, controlled trial (SB or placebo), with two arms parallel, randomized design, carried out on outpatient clinic because of acute bloody diarrhea.

DETAILED DESCRIPTION:
Patients with acute bloody diarrhea were prescribed randomly and blindly placebo or Saccharomyces boulardii 500 mg /day seven days (250 mg for children between 0.25 - 1.00 years),and were seen in outpatient clinics of three hospitals at days 1, 3, and 7. On day 14 they were contacted by telephone call. Parents registered daily number of stools, with or without diarrhea, and any new symptom appearing during follow up.

ELIGIBILITY:
Inclusion Criteria:

* all children between 0.25 and 5.99 years
* attending emergency clinic because of acute diarrhea,
* showing stools with presence of blood,
* whose parents were adequately informed, and signed the corresponding consent

Exclusion Criteria:

* diarrhea lasting more than 7 days at inclusion
* presence of malnutrition and any other chronic or major disease,
* previous or concomitant intake of steroids, or other immunosuppressive drugs,
* immunocompromised

Ages: 3 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2019-01-30 (Actual); Primary Completion 2026-01-26 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Duration of bloody diarrhea | From baseline to end of follow-up (Day 14)
  The number of days of bloody diarrhea between SB and placebo groups
Number of total stools per day | From baseline to end of follow-up (Day 14)
  Number of stools in children with or without blood in stools
Number of bloody stools per day | From baseline to end of follow-up (Day 14)
  Number of stools in children with blood in stools

SECONDARY OUTCOMES:
Proportion of patients with positive stool culture, ELISA, PCR | At baseline
  Stool culture for O157:H7 or non-O157:H7 enterohemorrhagic E. coli, PCR and/or ELISA for verotoxins and detection of Campylobacter spp, Shigella spp, Salmonella spp and other pathogens
Safety adverse events | From baseline to end of follow-up (Day 14)
  Differences in adverse events between both groups

CONTACTS AND LOCATIONS:
Overall Officials: Maria Gracia Caletti, Dr, Study Director; Diana Kelmansky, Dr, Principal Investigator — Statistician
Locations (3):
- Argentina (3):
  - Hospital Tetamanti in Mar del Plata (HIEMI), Mar del Plata, Buenos Aires
  - Hospital Ramos Mejía, Servicio de Pediatría (SPHRM), Buenos Aires, Buenos Aires F.D.
  - Hospital Materno Infantil de Salta, Salta, Salta Province

IPD SHARING:
Plan to Share IPD: Undecided